CLINICAL TRIAL: NCT01956942
Title: Phase IV Study of Micropulse Laser Trabeculoplasty Versus Selective Laser Trabeculoplasty for Treatment of Open Angle Glaucoma
Brief Title: Micropulse Laser Trabeculoplasty (MLT) Versus Selective Laser Trabeculoplasty (SLT) for Treatment of Open Angle Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Belyea (Other)
Responsible Party: Sponsor-Investigator, David Belyea, Principal Investigator, George Washington University
Organization: George Washington University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 041310
Record Dates: First submitted 2013-09-30; First posted 2013-10-08 (Estimated); Results first posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-05

CONDITIONS: Open Angle Glaucoma
Keywords: GLAUCOMA; MICROPULSE; LASER; TRABECULOPLASTY; OPEN ANGLE; INTRAOCULAR PRESSURE
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma | interventions — Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Micropulse Laser Trabeculoplasty (Experimental): Patient's randomized to MLT would be treated with the following settings: 300 micron spot size, 0.3 second duration, 15% duty cycle, and 1000 milliWatt power. They would be treated with confluent laser spots across the entire 360 degrees of the trabecular meshwork. Each patient would receive pre-treatment with a drop on iopidine or brimonidine to prevent post-operative intraocular pressure (IOP) spikes as per standard pre-laser trabeculoplasty protocol.
  Interventions: Device: Micropulse Laser Trabeculoplasty
- Selective Laser Trabeculoplasty (SLT) (Active Comparator): Patient's randomized to SLT would be treated with the following settings: 400 micron spot size, 0.3 second duration, and 1.00 milliWatt (mW) power. They would be treated with confluent laser spots across the entire 360 degrees of the trabecular meshwork. Each patient would receive pre-treatment with a drop on iopidine or brimonidine to prevent post-operative IOP spikes as per standard pre-laser trabeculoplasty protocol.
  Interventions: Device: Selective Laser Trabeculoplasty

INTERVENTIONS:
Device: Micropulse Laser Trabeculoplasty
  Other Names: MLT; Laser
  Arms: Micropulse Laser Trabeculoplasty
Device: Selective Laser Trabeculoplasty
  Other Names: SLT; Laser
  Arms: Selective Laser Trabeculoplasty (SLT)

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a new laser (called Micropulse Laser Trabeculoplasty or MLT) in the treatment of glaucoma compared to the conventional laser presently used which is called selective laser trabeculoplasty or SLT. Both lasers (SLT and MLT) are used as standard of care in the treatment of open angle glaucoma.

DETAILED DESCRIPTION:
Glaucoma is the 2nd leading cause of blindness worldwide and affects over 2.5 million Americans over the age of 40. It is thought that elevated intraocular pressure causes damage to the optic nerve fibers which leads to silent vision loss in glaucoma. Therefore, the primary approach to managing this disease process is through intraocular pressure reduction with a) topical drops that decrease intraocular fluid production or increase fluid outflow, b) laser therapy to the outflow structures in the eye (trabecular meshwork) to increase fluid egression, c) or incisional surgery with or without placement of setons to create a new pathway for fluid outflow. When medical therapy has been maximized or patients do not tolerate topical therapy, laser trabeculoplasty is common applied to achieve further intraocular pressure reduction. There are two types of laser therapies: argon laser trabeculoplasty (ALT) and selective laser trabeculoplasty (SLT). The former involves applying laser to create outflow pathways in the trabecular meshwork (TM) and induces thermal damage to the TM. The latter selectively applies energy which induces inflammatory restructuring of the TM without creating a burn. Studies have shown comparable results between the two treatment modalities with SLT offering the advantage of repeatable treatment. Studies have also shown laser trabeculoplasty to be comparable to the effect of topical drops in intraocular pressure reduction. Side effects for both types of laser trabeculoplasty include post procedure intraocular pressure elevation and intraocular inflammation which is treated with topical drops after the procedure.

This study aims to evaluate the effectiveness of micropulse laser trabeculoplasty in intraocular pressure reduction in patients with open angle glaucoma as compared to conventional selective laser trabeculoplasty. Secondary aims would be to determine whether its reduction is comparable to that of topical intraocular pressure lowering drops, length of therapeutic intraocular pressure reduction, and incidence of side effects commonly encountered with traditional laser trabeculoplasty including intraocular inflammation and intraocular pressure spikes.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any ange age
* Diagnosis of open angle glaucoma who have not had recent changes in their medication regimen.

Exclusion Criteria:

* Patients with active neovascularization of the angle, angle closure glaucoma, angle recession, or anterior uveitis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-08; Primary Completion 2017-07 (Actual); Study Completion 2017-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Belyea, MD, Principal Investigator — George Washington University
Locations (1):
- George Washington University Medical Faculty Associates, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Detry-Morel M, Muschart F, Pourjavan S. Micropulse diode laser (810 nm) versus argon laser trabeculoplasty in the treatment of open-angle glaucoma: comparative short-term safety and efficacy profile. Bull Soc Belge Ophtalmol. 2008;(308):21-8. PMID 18700451
- [Background] Juzych MS, Chopra V, Banitt MR, Hughes BA, Kim C, Goulas MT, Shin DH. Comparison of long-term outcomes of selective laser trabeculoplasty versus argon laser trabeculoplasty in open-angle glaucoma. Ophthalmology. 2004 Oct;111(10):1853-9. doi: 10.1016/j.ophtha.2004.04.030. PMID 15465546
- [Background] Fea AM, Bosone A, Rolle T, Brogliatti B, Grignolo FM. Micropulse diode laser trabeculoplasty (MDLT): A phase II clinical study with 12 months follow-up. Clin Ophthalmol. 2008 Jun;2(2):247-52. doi: 10.2147/opth.s2303. PMID 19668712

RESULTS

PARTICIPANT FLOW:
Groups:
- Micropulse Laser Trabeculoplasty: Patient's randomized to MLT would be treated with the following settings: 300 micron spot size, 0.3 second duration, 15% duty cycle, and 1000 milliWatt power. They would be treated with confluent laser spots across the entire 360 degrees of the trabecular meshwork. Each patient would receive pre-treatment with a drop on iopidine or brimonidine to prevent post-operative intraocular pressure (IOP) spikes as per standard pre-laser trabeculoplasty protocol.
  Micropulse Laser Trabeculoplasty
- Selective Laser Trabeculoplasty (SLT): Patient's randomized to SLT would be treated with the following settings: 400 micron spot size, 0.3 second duration, and 1.00 milliWatt (mW) power. They would be treated with confluent laser spots across the entire 360 degrees of the trabecular meshwork. Each patient would receive pre-treatment with a drop on iopidine or brimonidine to prevent post-operative IOP spikes as per standard pre-laser trabeculoplasty protocol.
  Selective Laser Trabeculoplasty
Period: Overall Study
Arm/Group | Micropulse Laser Trabeculoplasty | Selective Laser Trabeculoplasty (SLT)
Started | 38 | 31
Completed | 38 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Micropulse Laser Trabeculoplasty | Selective Laser Trabeculoplasty (SLT) | Total
Number analyzed (Participants) | 38 | 31 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 12 | 32
  >=65 years | 18 | 19 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.1 (0.3) | 67.6 (.85) | 66.9 (0.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 35
  Male | 22 | 12 | 34
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 38 | 31 | 69

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure Reduction
Description: evaluate the effectiveness of micropulse laser trabeculoplasty in intraocular pressure reduction in patients with open angle glaucoma as compared to conventional selective laser trabeculoplasty
  The aim of this study was to prospectively compare the efficacy, safety, and tolerability of selective laser trabeculoplasty (SLT) vs micropulse laser trabeculoplasty (MLT) in reducing intraocular pressure (IOP) in open-angle glaucoma patients.
Time Frame: within 6 weeks to 3 months after the laser procedure is completed
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Micropulse Laser Trabeculoplasty | Selective Laser Trabeculoplasty (SLT)
Number analyzed (Participants) | 38 | 31
percentage change | 17.01 (1) | 14.29 (1)

2. Primary Outcome: Intraocular Pressure (IOP) Reduction Comparison Between MLT and SLT
Description: Intraocular pressure (IOP) reduction comparison between MLT and SLT
Time Frame: 24-52 week interval
Population: A total of 69 patients with uncontrolled open-angle glaucoma were recruited, candidates with open-angle glaucoma on maximally tolerated medical therapy with the need for additional IOP lowering. All patients had only one eye included in the study.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Micropulse Laser Trabeculoplasty Group: Micropulse Laser Trabeculoplasty Group Treated
- Selective Laser Trabecuplasty Group: Selective Laser Trabeculoplasty Group
Arm/Group | Micropulse Laser Trabeculoplasty Group | Selective Laser Trabecuplasty Group
Number analyzed (Participants) | 38 | 31
mmHg | 15.7 (0.2) | 14.35 (0.3)

3. Primary Outcome: Intraocular Pressure (IOP) Reduction
Description: Percentage of participants with a decrease of greater or equal to 3 mmHg intraocular pressure from baseline
Time Frame: 52 weeks
Measure: Number; unit: percentage of participants
Groups:
- Selective Laser Trabeculoplasty Group: Selective Laser Trabeculoplasty Group
Arm/Group | Micropulse Laser Trabeculoplasty Group | Selective Laser Trabeculoplasty Group
Number analyzed (Participants) | 38 | 31
percentage of participants | 37 | 36

4. Secondary Outcome: Measurement of Pain/Inflammation by a Pain Scale Post Laser Treatments From Micropulse and Selective Laser Trabeculoplasty.
Description: The measurement of pain commonly encountered with traditional laser trabeculoplasty including intraocular inflammation will be measured and compared between both lasers (SLT vs. MLT).
  Standardized pain survey (scale of 0=none and 10=severe) Higher number, the more pain was being experienced by subject
Time Frame: at the time of treatment and at 1 week following the laser procedure
Measure: Mean (99% Confidence Interval); unit: score on a scale
Arm/Group | Micropulse Laser Trabeculoplasty Group | Selective Laser Trabecuplasty Group
Number analyzed (Participants) | 38 | 31
score on a scale
  During Treatment | 1.34 [0 to 10] | 2.83 [0 to 10]
  1 Week Post Treatment | 0.89 [0 to 10] | 2.81 [0 to 10]

ADVERSE EVENTS:
Time Frame: 52 weeks
Groups:
- Micropulse Laser Trabeculoplasty (MLT): Patient's randomized to MLT would be treated with the following settings: 300 micron spot size, 0.3 second duration, 15% duty cycle, and 1000 milliWatt power. They would be treated with confluent laser spots across the entire 360 degrees of the trabecular meshwork. Each patient would receive pre-treatment with a drop on iopidine or brimonidine to prevent post-operative intraocular pressure (IOP) spikes as per standard pre-laser trabeculoplasty protocol.
  Micropulse Laser Trabeculoplasty
Arm/Group | Micropulse Laser Trabeculoplasty (MLT) | Selective Laser Trabeculoplasty (SLT)
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/31
Other Adverse Events (participants affected / at risk) | 0/38 | 0/31

LIMITATIONS AND CAVEATS:
One site.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT01956942/Prot_SAP_000.pdf